CLINICAL TRIAL: NCT04789291
Title: A Randomised, Open-label, Single-dose, Two-way Cross-over Relative Bioavailability Comparison of BI 1595043 as Tablets With and Without Food in Healthy Male Subjects
Brief Title: A Study in Healthy Men to Test How BI 1595043 is Taken up in the Body When Given With or Without Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1445-0011; 2020-004924-40 (EudraCT Number)
Record Dates: First submitted 2021-03-08; First posted 2021-03-09 (Actual); Results first posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2023-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 1595043 fasted (Reference (R)) / BI 1595043 fed (Test (T)) (Experimental): Two period crossover separated by a wash-out of at least 8 days:
  Period 1: Healthy subjects received a single dose of 30 milligram (mg) BI 1595043 as film coated tablets (1x 5mg tablet and 1x 25mg tablet) following an overnight fast of at least 10 hours.
  Period 2: Healthy subjects received a single dose of 30 milligram (mg) BI 1595043 as film coated tablets (1x 5mg tablet and 1x 25mg tablet) following an following a high fat/high calorie breakfast.
  Interventions: Drug: BI 1595043
- BI 1595043 fed (Test (T)) / BI 1595043 fasted (Reference (R)) (Experimental): Two period crossover separated by a wash-out of at least 8 days:
  Period 1: Healthy subjects received a single dose of 30 milligram (mg) BI 1595043 as film coated tablets (1x 5mg tablet and 1x 25mg tablet) following an following a high fat/high calorie breakfast.
  Period 2: Healthy subjects received a single dose of 30 milligram (mg) BI 1595043 as film coated tablets (1x 5mg tablet and 1x 25mg tablet) following an overnight fast of at least 10 hours.
  Interventions: Drug: BI 1595043

INTERVENTIONS:
Drug: BI 1595043 — Single dose of 30 milligram (mg) BI 1595043 as film coated tablets (1x 5mg tablet and 1x 25mg tablet).

SUMMARY:
The main objective of this trial is to investigate the relative bioavailability of BI 1595043 under fed state (Test, T) and under fasted state (Reference, R).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR), body temperature), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation
* Male subjects who meet any of the following criteria from at least 30 days before the first administration of trial medication until 30 days after trial completion:

  * Use of adequate contraception, i.e. use of condom (male subjects) plus any of the following methods (female partners): intrauterine device, hormonal contraception (e.g. implants, injectables, combined oral or vaginal contraceptives) that started at least 2 months prior to first drug administration to the male subject, or barrier method (e.g. diaphragm with spermicide), or surgically sterilised (including bilateral tubal occlusion, hysterectomy or bilateral oophorectomy), or postmenopausal, defined as at least 1 year of spontaneous amenorrhea
  * Sexually abstinent
  * Vasectomised (vasectomy at least 1 year prior to enrolment) in combination with a barrier method (i.e. condom) Unprotected sexual intercourse (i.e. without use of condom) with a pregnant female partner and sperm donation is not allowed throughout the study and until 30 days after trial completion

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2021-08-07 (Actual); Study Completion 2021-08-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, randomised, single centre trial using a two-way cross-over design. All subjects received a single oral dose of 30 mg BI 1595043 in film-coated tablet formulation following an overnight fast and after the ingestion of a standardised, high-calorie, high-fat breakfast. Administration sequence was randomly allocated with a wash-out period of at least 8 days between BI 1595043 doses.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Period 1
Arm/Group | BI 1595043 Fasted (Reference (R)) / BI 1595043 Fed (Test (T)) | BI 1595043 Fed (Test (T)) / BI 1595043 Fasted (Reference (R))
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0
Period: Wash-out
Arm/Group | BI 1595043 Fasted (Reference (R)) / BI 1595043 Fed (Test (T)) | BI 1595043 Fed (Test (T)) / BI 1595043 Fasted (Reference (R))
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0
Period: Period 2
Arm/Group | BI 1595043 Fasted (Reference (R)) / BI 1595043 Fed (Test (T)) | BI 1595043 Fed (Test (T)) / BI 1595043 Fasted (Reference (R))
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): included all subjects who were randomised and received at least one dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 1595043 Fasted (Reference (R)) / BI 1595043 Fed (Test (T)) | BI 1595043 Fed (Test (T)) / BI 1595043 Fasted (Reference (R)) | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (7.9) | 38.2 (5.8) | 35.5 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 1595043 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of BI 1595043 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) is reported.
  The statistical model used was an analysis of variance (ANOVA) model on the logarithmic scale. Data was logtransformed (natural logarithm) prior to fitting the ANOVA model.This model included effects accounting for the following sources of variation: 'sequence', 'subjects within sequences', 'period' and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed.
Time Frame: Within 3 hours before drug administration and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 34, 48, 72, 96, 120, 144 and 168 hours following drug administration.
Population: Pharmacokinetic parameter analysis set (PKS): all subjects who were randomised and received at least one dose of trial medication and who provided at least one pharmacokinetic (PK) endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Standard Error); unit: hour*nanomol/Liter
Groups:
- BI 1595043 Under Fasted Condition (Reference (R)): Healthy subjects received a single dose of 30 milligram (mg) BI 1595043 as film coated tablets (1x 5mg tablet and 1x 25mg tablet) following an overnight fast of at least 10 hours.
- BI 1595043 Under Fed Condition (T (Test)): Healthy subjects received a single dose of 30 milligram (mg) BI 1595043 as film coated tablets (1x 5mg tablet and 1x 25mg tablet) following an following a high fat/high calorie breakfast.
Arm/Group | BI 1595043 Under Fasted Condition (Reference (R)) | BI 1595043 Under Fed Condition (T (Test))
Number analyzed (Participants) | 13 | 13
hour*nanomol/Liter | NA (NA) — Geometric Mean is actually adjusted Geometric Mean = 4130.12. Standard Error is actually adjusted Geometric Standard Error = 1.06. | NA (NA) — Geometric Mean is actually adjusted Geometric Mean = 4244.02. Standard Error is actually adjusted Geometric Standard Error = 1.06.
Statistical Analysis 1: Comparison: BI 1595043 Under Fasted Condition (Reference (R)) vs BI 1595043 Under Fed Condition (T (Test)); Relative bioavailability of BI 1595043 administered in fed state (Test) compared with BI 1595043 administered in fasted state (Reference) was estimated by the ratios of the gMeans (Test/Reference). Their corresponding 2-sided 90% CIs were provided. This method corresponds to 2 one-sided t-test procedures, each at the 5% significance level; Test type: Other; Ratios of adjusted geometric means [%] = 102.76, 90% CI 2-sided [99.34 to 106.29] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 4.8

2. Primary Outcome: Maximum Measured Concentration of BI 1595043 in Plasma (Cmax)
Description: Maximum measured concentration of BI 1595043 in plasma (Cmax) is reported.
  The statistical model used was an analysis of variance (ANOVA) model on the logarithmic scale. Data was logtransformed (natural logarithm) prior to fitting the ANOVA model.This model included effects accounting for the following sources of variation: 'sequence', 'subjects within sequences', 'period' and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: nanomol/Liter
Groups:
- Reference (R) BI 1595043 Under Fasted Condition: Healthy subjects received a single dose of 30 milligram (mg) BI 1595043 as film coated tablets (1x 5mg tablet and 1x 25mg tablet) following an overnight fast of at least 10 hours.
- T (Test) BI 1595043 Under Fed Condition: Healthy subjects received a single dose of 30 milligram (mg) BI 1595043 as film coated tablets (1x 5mg tablet and 1x 25mg tablet) following an following a high fat/high calorie breakfast.
Arm/Group | Reference (R) BI 1595043 Under Fasted Condition | T (Test) BI 1595043 Under Fed Condition
Number analyzed (Participants) | 13 | 13
nanomol/Liter | NA (NA) — Geometric Mean is actually adjusted Geometric Mean = 810.95. Standard Error is actually adjusted Geometric Standard Error = 1.06. | NA (NA) — Geometric Mean is actually adjusted Geometric Mean = 630.96. Standard Error is actually adjusted Geometric Standard Error = 1.06.
Statistical Analysis 1: Comparison: Reference (R) BI 1595043 Under Fasted Condition vs T (Test) BI 1595043 Under Fed Condition; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratios of adjusted geometric means [%] = 77.81, 90% CI 2-sided [69.77 to 86.76] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 15.5

3. Secondary Outcome: Area Under the Concentration-time Curve of BI 1595043 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of BI 1595043 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is reported.
  The statistical model used was an analysis of variance (ANOVA) model on the logarithmic scale. Data was logtransformed (natural logarithm) prior to fitting the ANOVA model.This model included effects accounting for the following sources of variation: 'sequence', 'subjects within sequences', 'period' and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: hour*nanomol/Liter
Arm/Group | Reference (R) BI 1595043 Under Fasted Condition | T (Test) BI 1595043 Under Fed Condition
Number analyzed (Participants) | 13 | 13
hour*nanomol/Liter | NA (NA) — Geometric Mean is actually adjusted Geometric Mean = 4191.59. Standard Error is actually adjusted Geometric Standard Error = 1.07. | NA (NA) — Geometric Mean is actually adjusted Geometric Mean = 4327.59. Standard Error is actually adjusted Geometric Standard Error = 1.07.
Statistical Analysis 1: Comparison: Reference (R) BI 1595043 Under Fasted Condition vs T (Test) BI 1595043 Under Fed Condition; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratios of adjusted geometric means [%] = 103.24, 90% CI 2-sided [99.73 to 106.89] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 4.9

ADVERSE EVENTS:
Time Frame: From the day of study drug administration till the next administration or until end of trial, whatever occurred first, up to 14 days.
Description: Treated set (TS): This analysis set included all subjects who were randomised and received at least one dose of trial medication.
Arm/Group | BI 1595043 Under Fed Condition (T (Test)) | BI 1595043 Under Fasted Condition (Reference (R))
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 1/13 | 2/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1595043 Under Fed Condition (T (Test)) (N=13) | BI 1595043 Under Fasted Condition (Reference (R)) (N=13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/91/NCT04789291/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/91/NCT04789291/SAP_001.pdf